CLINICAL TRIAL: NCT03309306
Title: Evaluating Household Food Behavior With a Smartphone App
Acronym: FoodImage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PBRC 2017-042
Record Dates: First submitted 2017-10-03; First posted 2017-10-13 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Food Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A subset of subjects will complete Phase I, which is the lab-based portion of the study, prior to the RCT.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: Lab Testing (Visit 1, Day 0) (No Intervention): In a laboratory kitchen, participants will use the following 3 methods to record and measure food waste during simulated shopping trip and kitchen clean-outs: the FoodImage App, Pen-and-paper Records, and Pen-and-paper records with a scale. Measurements will be collected by participants with all three methods, while lab personnel directly weigh foods to provide the criterion value.
- Phase 2: RCT Stress Management (Active Comparator): Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges in free-living conditions. Participants will capture baseline data for 4-7 days. After a 1-week break, participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also receive information on stress management
  Interventions: Other: Natural Environment/Stress Management
- Phase 2: RCT Food Waste Reduction (Experimental): Phase 2 will occur in participants' natural environment (free-living conditions). Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges. Participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also be provided with the following:
  1. Feedback on the amount of food waste their household created during the first week,
  2. A goal to reduce the next week's food waste by 20% or more, and
  3. Tips on how to reduce household food waste adapted from current consumer campaigns
  Interventions: Behavioral: Natural Environment/Reduce Food Waste

INTERVENTIONS:
Other: Natural Environment/Stress Management — Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges in free-living conditions. Participants will capture baseline data for 4-7 days. After a 1-week break, participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also receive information on stress management
  Arms: Phase 2: RCT Stress Management
Behavioral: Natural Environment/Reduce Food Waste — Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges in free-living conditions. Participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also be provided with the following:
  1. Feedback on the amount of food waste their household created during the first week,
  2. A goal to reduce the next week's food waste by 20% or more, and
  3. Tips on how to reduce household food waste adapted from current consumer campaigns
  Arms: Phase 2: RCT Food Waste Reduction

SUMMARY:
The purpose of this study is to test the use of a smartphone app as a way to measure food waste.

Investigators propose to improve the accuracy and convenience of household food waste measurement so that consumer food waste program evaluations yield more power, less bias, less measurement error, and greater representation of targeted populations.

DETAILED DESCRIPTION:
Investigators will improve measurement via the development of the FoodImage smartphone app, a technology leveraging the investigators' expertise in creating and deploying apps to measure food intake and deliver nutritional interventions in free-living household conditions. Investigators will validate the app against weighed waste in a controlled laboratory setting.

The study will yield an app ready for future study deployment while analyses of the data will inform rapidly evolving policy discussions concerning optimal approaches to reduce food waste. These outcomes align with program priorities to understand the economics of food waste and to use behavioral economics to address consumption behavior.

Specific objectives include:

1. Development of FoodImage, a smartphone app that measures household food waste and food-waste-related behaviors,
2. Assess differences in the accuracy and time burden of measurements taken with the FoodImage app versus two current household food waste measurement approaches (a pen-and-paper diary, and a pen-and-paper diary with a scale).
3. Use the FoodImage app in a pilot randomized controlled trial designed to evaluate the effectiveness of reducing household food waste through behavioral nudges in the form of personalized feedback about food waste levels and household-specific reduction goals.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* body mass index 18.5 - 50 kg/m2, based on self-reported height and weight
* Shops for groceries
* Conducts some of the food shopping and food preparation for their household
* Be willing to do food shopping for the study (if necessary)
* Have an iPhone and an operable Apple ID, password, and email address and is willing to use these to collect data during the study, acknowledging that data usage, and associated charges, are a result of study participation
* Be willing to complete all study procedures corresponding to their randomization group

Exclusion Criteria:

In addition to those who do not meet inclusion criteria, subjects who meet any of the following criteria will be excluded from enrollment:

* Persons who are severely immune compromised
* Persons who are pregnant, as assessed by self-report
* Pennington employee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roe BE, Qi D, Beyl RA, Neubig KE, Martin CK, Apolzan JW. The Validity, Time Burden, and User Satisfaction of the FoodImage Smartphone App for Food Waste Measurement Versus Diaries: A Randomized Crossover Trial. Resour Conserv Recycl. 2020 Sep;160:104858. doi: 10.1016/j.resconrec.2020.104858. Epub 2020 May 21. PMID 32773964

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: RCT Food Waste Reduction: Phase 2 will occur in participants' natural environment (free-living conditions). Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges. Participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also be provided with the following:
  1. Feedback on the amount of food waste their household created during the first week,
  2. A goal to reduce the next week's food waste by 20% or more, and
  3. Tips on how to reduce household food waste adapted from current consumer campaigns
  Natural Environment/Reduce Food Waste: Participants will use the FoodImage app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from food purges in free-living conditions. Participants will use the app to record food waste for approximately 4-7 days over the subsequent week. They will also be provided with the following:
  1. Feedback on the amount of food waste their household created during the first week,
  2. A goal to reduce the next week's food waste by 20% or more, and
  3. Tips on how to reduce household food waste adapted from current consumer campaigns
Period: Overall Study
Arm/Group | Phase 2: RCT Stress Management | Phase 2: RCT Food Waste Reduction
Started (Two participants dropped out of the study during the baseline assessment period, prior to being randomized to treatment) | 23 | 19
Completed | 22 | 18
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Includes individuals recruited to participate, screened for eligibility, and measured at baseline. Arms/Groups are combined because baseline measures were collected prior to randomization.
Groups:
- All Participants: All individuals recruited to participate in the study. Arms/Groups are combined because baseline measures were collected prior to randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 36.3 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Avoidable waste [Mean (Standard Deviation); unit: grams/week] | 741.5 (984.4)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Food Waste Error
Description: Participant estimations of food waste using the following three experimental methods as compared to the criterion value of weighed waste collected by study staff: 1) the FoodImage App (FoodImage app estimates minus the criterion value of lab personnel measured weighed food waste), 2) pen and paper diary with visual estimation of food amounts (pen and paper estimates minus the criterion value), and 3) pen and paper diary with a scale (pen and paper dairy accompanied by a scale minus directly weighed foods by lab personnel). All food values are in grams. The error values noted here represent less accurate estimates the further away they are from zero, either in the positive or negative direction. There are no min and max values to error measures.
Time Frame: Visit 1
Measure: Mean (Standard Deviation); unit: grams
Groups:
- FoodImage App: Participants will use the FoodImage app to measure food waste during simulated shopping trip and kitchen clean-out. Measurements will be collected by participants while lab personnel directly weigh foods to provide the criterion value.
- Diary: Visual Estimation: Participants will use pen and paper food records to measure food waste during simulated shopping trip and kitchen clean-out. Measurements will be collected by participants while lab personnel directly weigh foods to provide the criterion value.
- Diary With a Scale: Participant estimated food waste where a pen and paper diary was used accompanied by a scale.
Arm/Group | FoodImage App | Diary: Visual Estimation | Diary With a Scale
Number analyzed (Participants) | 23 | 23 | 23
grams | -16.25 (84.72) | 31.34 (134.80) | 20553.6 (111,151)

2. Secondary Outcome: Phase 2: Weight of All Household Waste
Description: Difference in change in total weight of all sources of household food waste.
Time Frame: Baseline to Day 14
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Phase 2: RCT Stress Management | Phase 2: RCT Food Waste Reduction
Number analyzed (Participants) | 22 | 18
grams | -232.65 (289.44) | -325.05 (319.99)

ADVERSE EVENTS:
Time Frame: 4 hours
Groups:
- All Participants: All individuals who completed the study
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT03309306/Prot_SAP_005.pdf